CLINICAL TRIAL: NCT02148848
Title: A Comparative Study of Short-term Functional Recovery Between Early- and Late Bisphosphonate Treatment Following Hemiarthroplasty in Patients With Osteoporotic Femoral Neck Fractures
Brief Title: Short-term Functional Recovery Between Early- and Late Bisphosphonate Treatment Following Hemiarthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 229/2556(EC4)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Osteoporotic Fractures; Femoral Neck Fracture
Keywords: Osteoporosis; Femoral neck fracture; hemiarthroplasty
MeSH Terms: conditions — Osteoporotic Fractures; Femoral Neck Fractures; Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early bisphosphonate use (Active Comparator): Give risedronate (actonel) at 2 weeks after hemiarthroplasty for an osteoporotic femoral neck fracture. In addition, calcium and vitamin D supplementation will be given to all patients.
  Risedronate (35 mg) 1 tablet orally once a week
  Interventions: Drug: Risedronate
- Late bisphosphonate use (No Intervention): Give only calcium and vitamin D supplementation during the first 3 months after the surgery.
  Bisphosphonate, risedronate (Actonel), will be given at 3 months after surgery for an osteoporotic femoral neck fracture.

INTERVENTIONS:
Drug: Risedronate — Take risedronate 35 mg orally every week
  Other Names: Actonel
  Arms: Early bisphosphonate use

SUMMARY:
Femoral neck fracture in the elderly is one indication for initiating osteoporosis treatment. Bisphosphonates remain the first line therapy; however, many orthopaedic surgeons concern regarding their effects on fracture healing process. Therefore, therapy is usually delayed for a period of time. To the best of our knowledge, there is no scientific data to support whether bisphosphonate treatment should be given immediately after the surgery or it should be delayed.

DETAILED DESCRIPTION:
Femoral neck fracture in the elderly is one indication for initiating osteoporosis treatment. Bisphosphonates remain the first line therapy; however, many orthopaedic surgeons concern regarding their effects on fracture healing process. Therefore, therapy is usually delayed for a period of time. To the best of our knowledge, there is no scientific data to support whether bisphosphonate treatment should be given immediately after the surgery or it should be delayed.

This study aims to compare functional recovery between early- and late administration of bisphosphonate in patients who received hemiarthroplasty following femoral neck fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with femoral neck fracture and was treated with bipolar hemiarthroplasty
* Age more than 50 years old and bone mineral density (BMD) was in osteoporotic (T-score less than -2.5) or osteopenic (T-score between -1.0 and -2.5) ranges

Exclusion Criteria:

* Patients who were treated with bipolar hemiarthroplasty for more than 2 weeks
* Patients with postoperative complications which affect the postoperative rehabilitation program e.g. intraoperative cracking or fracture, postoperative cardiac complication
* Have contraindications for bisphosphonates use e.g. renal insufficiency (glomerular filtration rate (GFR) < 30 ml/min), allergy to bisphosphonates, severe esophagitis, gastroesophageal reflux disease etc.
* Patients with conditions/disorders which have an affect on bone mineral density or bone metabolism e.g. renal insufficiency, rheumatoid arthritis, Paget's disease, renal osteodystrophy, hyperparathyroidism, glucocorticoids use etc.
* History of bisphosphonates use within 12 months
* Open fracture, multiple fracture or multiple trauma patients
* Pathological fracture
* Bilateral lower extremity fractures
* The pre-injury functional status of the patients is non-ambulatory

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
de Morton Mobility Index | 3 months after surgery

SECONDARY OUTCOMES:
Barthel index | 3 months after surgery
Visual analog scale score | 3 months after surgery
Two minutes walking test | 3 months after surgery
Timed get up and go test | 3 months after surgery
EuroQoL-5D (EQ-5D) | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aasis Unnanuntana, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Derived] Unnanuntana A, Laohaprasitiporn P, Jarusriwanna A. Effect of bisphosphonate initiation at week 2 versus week 12 on short-term functional recovery after femoral neck fracture: a randomized controlled trial. Arch Osteoporos. 2017 Dec;12(1):27. doi: 10.1007/s11657-017-0321-8. Epub 2017 Mar 10. PMID 28283937